CLINICAL TRIAL: NCT06829992
Title: Effects of Applying Kinesio Tapping on Primary Dysmenorrhea in Football Players: Randomized Clinical Trial
Brief Title: Effects of Applying Kinesio Tapping on Primary Dysmenorrhea in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Maíta Poli de Araújo, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 6665758; 76907423.1.0000.5505 (Registry Identifier: 76907423.1.0000.5505)
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Primary Dysmenorrhea (PD)
Keywords: primary dysmenorrhea; kinesio taping; female football

STUDY DESIGN:
Intervention Model Description: Kinesio Taping group and placebo group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Kinesio Taping group (Experimental): KT will be applied by a physiotherapist with experience in the Kinesio Taping method by Kenzo Kase.
  Three I-shaped Kinesio tapes will be used, 5 cm wide, covering the T-11 and T-12 dermatomes.
  The first tape will be applied vertically between the navel and pubis, with the participant in an orthostatic position with slight trunk extension. The second tape, with the same length as the first, will be applied with its central region over the middle zone of the first, perpendicularly. The third tape will be applied horizontally to the lower back, covering the spines posterosuperior iliac muscles, with the participant in an orthostatic position, performing light trunk flexion.
  Interventions: Device: Kinesio Taping
- placebo group (Placebo Comparator): The quantity of tapes, type, size and region of application will be the same as the group KT, however, in this group the tapes will be applied without tension and with procedure different from that recommended, first starting to adhere a side anchor into the skin, followed by the center and then the other side anchor.
  Interventions: Device: Placebo Group

INTERVENTIONS:
Device: Kinesio Taping — KT will be applied by a physiotherapist with experience in the Kinesio Taping method by Kenzo Kase. Three I-shaped Kinesio tapes will be used, 5 cm wide, covering the T-11 and T-12 dermatomes. The first tape will be applied vertically between the navel and pubis, with the participant in an orthostatic position with slight trunk extension.
  The second tape, with the same length as the first, will be applied with its central region over the middle zone of the first, perpendicularly. The third tape will be applied horizontally to the lower back, covering the spines posterosuperior iliac muscles, with the participant in an orthostatic position, performing light trunk flexion.
  Other Names: Taping; Tape
  Arms: Kinesio Taping group
Device: Placebo Group — The quantity of tapes, type, size and region of application will be the same as the group KT, however, in this group the tapes will be applied without tension and with procedure different from that recommended, first starting to adhere a side anchor into the skin, followed by the center and then the other side anchor.
  Other Names: placebo
  Arms: placebo group

SUMMARY:
The objective of this clinical study is to investigate the effects of applying Kinesio Taping to female soccer players with PD and comparing this application with a placebo group.

DETAILED DESCRIPTION:
Women's football has grown in the last decade, but there is still a need to study how the menstrual cycle affects players' performance. Primary Dysmenorrhea (PD), a common menstrual pain, impacts between 50% and 90% of women, reducing their participation in sporting activities. Many players notice that their performance is affected during the cycle, and the use of anti-inflammatories is not always effective. Therefore, it is important to implement simple measures that improve the quality of life and performance of players. Alternatives such as physical therapy and Kinesio Taping (KT) can help alleviate symptoms. The literature shows that KT is a technique with the potential to produce tactile sensory impulses on the skin, which can block or reduce the arrival of painful sensations to the brain, and could therefore be interesting in the treatment of PD. Therefore, the present study aims to investigate the effects of applying Kinesio Taping to female soccer players with PD and comparing this application with a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Women practicing football from the Mulheres em Campo project
* Primary dysmenorrhea
* Aged between 15 and 17 years
* Regular menstrual cycle (28 ± 7 days)
* Nulliparous
* Not having an intrauterine contraceptive device or using oral contraceptives
* DP will be defined according to the Visual Analogue Scale from 5 points.

Exclusion Criteria:

* Women who do not play football in the Mulheres em Campo project
* Secondary dysmenorrhea
* Diagnosed with serious comorbidity
* Skin lesions in the abdominal region
* Allergy to adhesive tapes.

Ages: 15 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Women
Enrollment: 50 (Actual)
Dates: Start 2025-05-26 (Actual); Primary Completion 2025-09-27 (Actual); Study Completion 2025-11-18 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | At recruitment and at the end of the menstrual cycle of each of the four months of the study (each cycle is 28 days).
  Visual Analogue Scale (VAS): to assess the intensity of menstrual pain. 10 cm VAS, which proved to be a valid and reliable tool for measuring experimental and clinical pain. The VAS is scored on a horizontal line of 10 points (0 = no pain and 10 = maximum pain). Participants must mark the intensity of menstrual pain on the horizontal line, considering the most painful days of the menstrual cycle.

SECONDARY OUTCOMES:
Short McGill | At recruitment and at the end of the menstrual cycle of each of the four months of the study (each cycle is 28 days)
  Assessment of subjective pain in relation to PD. Shortened version of the original McGill questionnaire, translated and validated into Portuguese. The person assessed must choose one of 15 words and the pain is classified according to its sensory and affective dimensions, along with an analogue scale that assesses the general intensity of the pain in the last few days and a 6-item scale with a global description of the intensity. The questionnaire score is calculated based on the intensity of the pain descriptors chosen by the patient. Being the intensity scale 0 = none, 1 = mild, 2 = uncomfortable, 3 = distressing, 4 = horrible, 5 = excruciating. The pain index is obtained by adding the intensity values of the chosen descriptors. The highest possible value is 20, as the patient can only choose one word per subgroup. The higher the total score, the greater the patient's pain experience.
Menstrual complaints questionnaire | At recruitment and at the end of the menstrual cycle of each of the four months of the study (each cycle is 28 days)
  Assessment of the presence of low back pain, headache, abdominal swelling, breast tenderness, fatigue, nausea, vomiting, diarrhea, constipation, insomnia, nervousness and depression. Responses will be recorded as "present" or "absent" on a questionnaire
Questionnaire on interference of Primary Dysmenorrhea in sports practice | At recruitment and at the end of the menstrual cycle of each of the four months of the study (each cycle is 28 days)
  Assessment of how much the symptoms of primary dysmenorrhea interfered with their sports practice. The responses will be recorded as "almost no interference", "little interference", "medium interference", "a lot of interference", "intense interference".
Short form health survey 36 (sf-36) | At recruitment and at the end of the menstrual cycle of each of the four months of the study (each cycle is 28 days)
  Assessment of quality of life. Translated and validated version into Portuguese of the Short Form Health Survey 36. The SF-36 assesses eight aspects of quality of life: Functional capacity, Physical aspects, Emotional aspects, Pain, General health status, Vitality, Social aspects, Mental health. Your score ranges from 0 to 100, with 0 being the worst health status and 100 being the best.
Diary menstrual | Every day of the menstrual cycle throughout the four months of the study (each cycle is 28 days)
  Paper diary where they must record with a pen every time they take medication due to discomfort related to dysmenorrhea in each menstrual cycle, as well as the intensity of the discomfort (mild, moderate, intense).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gynecology of Federal University of São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be authorized because the sample is made up of minors and the information collected is confidential. After the study is completed, the results will be duly published in accordance with ethical standards.